CLINICAL TRIAL: NCT01472861
Title: A Randomized Controlled Trial Evaluating Autologous Endometrial Coculture (AECC) As An Effective Tool For Young Patients With Poor Ovarian Reserve
Brief Title: Autologous Endometrial Coculture (AECCT)
Acronym: AECCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0903010293
Record Dates: First submitted 2011-11-11; First posted 2011-11-17 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Infertility
Keywords: coculture; endometrial biopsy; IVF poor responders
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No AECC (Placebo Comparator): Routine procedures without AECC
  Interventions: Other: no endometrial biopsy or Autologous endometrial coculture (AECC) performed
- AECC (Experimental): Endometrial biopsy and Autologous endometrial coculture
  Interventions: Procedure: AECC (Autologous endometrial coculture)

INTERVENTIONS:
Procedure: AECC (Autologous endometrial coculture) — endometrial biopsy with autologous endometrial coculture
  Arms: AECC
Other: no endometrial biopsy or Autologous endometrial coculture (AECC) performed — routine procedures with out biopsy
  Arms: No AECC

SUMMARY:
The purpose of this study is to determine if the use of Autologous Endometrial Coculture (AECC) in young in vitro fertilization (IVF) patients with poor ovarian reserve improves pregnancy outcome.

DETAILED DESCRIPTION:
Young women with poor ovarian reserve are commonly given a poor prognosis for IVF success. Standard culture media for fertilizing oocytes (unfertilized eggs) is commonly used in IVF which closely resembles tubal fluid. Efforts to create optimal culture conditions for fertilization of human embryos for women with poor quality embryos and/or repeated implantation failures have been developed at our center by using AECC. AECC involves placing a patient's fertilized eggs on top of a layer of cells from her own uterine lining, creating a more natural environment for embryo development and maximizing the chance for IVF pregnancy. The investigators will prospectively randomize young patients (≤ age 38 years) poor ovarian reserve to AECC or no AECC with standard culture media to study pregnancy outcome.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women undergoing IVF at CRMI
* Age ≤ 38 years
* Poor ovarian reserve with antral follicle count less than 6 follicles, cycle day 2/3 FSH > 12 ng/ml, AMH < 0.5 ng/ml

Exclusion Criteria:

* Healthy women undergoing IVF with male factor, severe endometriosis, or tubal factor infertility
* Donor patients
* Contraindications for the use of gonadotropins (i.e. pregnancy, lactation, undiagnosed vaginal bleeding or ovarian cysts)
* Recent or current medical conditions where the patient is not medically stable to undergo stimulation or egg retrieval, HIV infection, diabetes, cardiovascular disease, gastrointestinal, hepatic disease, renal or pulmonary disease.
* Any patient who is not a candidate for IVF

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pregnancy outcome | 1 month

SECONDARY OUTCOMES:
Embryo quality | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Spandorfer Steven, MD, Principal Investigator — Weill Medical College
Locations (1):
- Center for Reproducutve Medicine; Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- See also: Ronald O. Perelman and Claudia Cohen Center for Reproductive Medicine — http://ivf.org